CLINICAL TRIAL: NCT01147913
Title: Computerized Information-Processing Bias Retraining in Adolescents With Depression: A Controlled Trial
Brief Title: Computerized Information-Processing Bias Retraining in Depressed Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jamie A. Micco, PhD, Assistant in Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F32MH088065-01
Record Dates: First submitted 2010-04-12; First posted 2010-06-22 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Major Depression
Keywords: Major Depression; Depression; Anxiety; Dysthymia
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Anxiety Disorders; Dysthymic Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive Interpretation Training (Experimental): Four sessions of positive information-processing training for interpretation of ambiguous scenarios relevant to themes of depression.
  Interventions: Behavioral: Computerized Information-Processing Bias Retraining
- Attention Control Training (Sham Comparator): Four sessions of interpretation training for "filler" or neutral scenarios, unrelated to themes associated with depression.
  Interventions: Behavioral: Attention Control Training

INTERVENTIONS:
Behavioral: Computerized Information-Processing Bias Retraining — The intervention consists of the presentation of three-line ambiguous scenarios via a computer program, one line at a time. A disambiguating word fragment completes the scenario (in either a positive or neutral valence, depending on the scenario), after which participants will type the first letter of the word on the keyboard to ensure they are encoding the interpretation valence. The computer will indicate if they have correctly identified the word. This is followed by a Y/N comprehension question. Each session presents 100 training scenarios.
  Arms: Positive Interpretation Training
Behavioral: Attention Control Training — Four sessions of interpretation training for "filler" or neutral scenarios, unrelated to themes associated with depression.
  Arms: Attention Control Training

SUMMARY:
This study will examine how well a novel four-session computerized program, designed to help adolescents learn to interpret ambiguous situations less negatively, reduces symptoms of depression and decreases negative information-processing biases.

DETAILED DESCRIPTION:
Major Depression is a markedly impairing disorder that affects up to 20% of adolescents before adulthood, and is associated with significant impairment in adolescents' emotional and social development. While antidepressant medication and psychotherapy are effective in treating some depressed adolescents, approximately 30% fail to respond to a combination of these treatments. Furthermore, many families are reluctant to pursue antidepressant medication for depressed adolescents because of concerns about potentially increasing risk of suicidal ideation. Thus, there is a critical need for effective, non-pharmacological treatments for this population. One promising new intervention consists of modifying negative information-processing biases associated with depression. Recent research has suggested that these biases may be modified using a computerized program that provides repeated exposure to positive interpretations of salient, ambiguous situations, with the goal of interpreting ambiguity less negatively. These modification programs have been efficacious in altering interpretation biases and reducing anxiety in adults with social and specific phobias. Therefore, the proposed study aims to examine the efficacy of an adapted interpretation bias modification program for depressed adolescents. Specifically, the study will examine the efficacy of four sessions of the modification program in altering interpretation biases and reducing symptoms of depression, anxiety, and negative affect. A total of 60 adolescents (ages 14-21) with symptoms of major depression will be randomly assigned to either the active intervention condition (four sessions of the modification program over two weeks) or an attention control condition. Measures will include a diagnostic interview, self-report measures of depression, anxiety, and negative affect, and a test of interpretation bias in response to ambiguous situations. It is hypothesized that: 1) Compared to adolescents in the attention control condition, adolescents who receive four sessions of the positive interpretive training will experience a significantly larger decrease from baseline to post-treatment in negative interpretation bias (e.g., more positive and fewer negative interpretations of ambiguous situations) on a measure of interpretation bias; and, 2)Compared to adolescents in the attention control condition, adolescents who receive the positive interpretation training will experience a significantly larger decrease from baseline to post-treatment in self-reported state depression, anxiety, and negative affect.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 14-21 years old
* A score of 14 or higher on the Beck Depression Inventory, 2nd Edition (BDI-II)
* Working command of the English language

Exclusion Criteria:

* Psychosis, current mania, or acute suicidality
* Previous diagnosis of pervasive developmental disorder, mental retardation, or severe dyslexia
* Changes in psychiatric medication or psychotherapy within two weeks of entering the study

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Test of Interpretation Bias (TIB) | up to 1 day post-treatment
  The TIB consists of 10 scenarios, similar to the training scenarios except that the last word of all of the scenarios remains ambiguous in valence. Following exposure to each of these ambiguous scenarios, adolescents are given a series of four statements regarding the scenario and asked to rate on a 4-point scale how similar the statement is to their interpretation of the scenario. Two target statements are presented, one with the positive interpretation and one with the negative interpretation. Scores for negative and positive interpretations across the situations can then be calculated.
Test of Interpretation Bias | 2-Week Follow-Up
  See above

SECONDARY OUTCOMES:
Kiddie-Schedule of Affective Disorders and Schizophrenia-Epidemiologic Version (K-SADS-E; Orvaschek & Puig-Antich, 1987) | up to one day Post-Treatment and at 2-Week Follow-Up
  DSM-IV structured interview for children up to age 16 years old; assesses for major depression, dysthymia, and mania.
Beck Depression Inventory, 2nd Version | up to 1 day Post-Treatment and at 2-Week Follow-Up
  The BDI-II is a questionnaire the measures symptoms of depression over the previous two weeks.
State-Trait Anxiety Scale (STAI) | up to 1 day Post-Treatment and 2-Week Follow-Up
  The STAI is a self-report measure of anxiety symptoms over the past week (trait) and currently (state).
Structured Clinical Interview for DSM-IV (SCID-IV; First et al, 1997), Mood Disorder Modules only | up to 1 day Post-Treatment and 2-Week Follow-Up
  DSM-IV structured interview for adults (17 years old and older); assesses for major depression, dysthymia, and mania
Dysfunctional Attitudes Scale (DAS) | up to 1 day post-treatment and at two-week follow-up
  The DAS-A is a 40-item self-report measure of depressogenic beliefs. The scale has two factors: Perfectionism and Need for Social Approval (Imber et al., 1990). Internal consistency and concurrent validity have been found to be acceptable (Imber et al, 1990; Blatt et al, 1995).
CANTAB Affective Go-No Go Task (AGN) | up to 1 day post-treatment
  The AGN test assesses information processing biases for positive and negative stimuli and takes 10 minutes to administer. The test consists of several blocks, each of which presents a series of words from two of three different Affective categories: Positive (for example, joyful), Negative (for example, hopeless), and Neutral (for example, element). The subject is given a target category, and is asked to press the press pad when they see a word matching this category. There are twelve outcome measures covering latency and errors of commission and omission.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie A Micco, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Clinical and Research Program in Pediatric Psychopharmacology at Massachusetts General Hospital, Cambridge, Massachusetts, United States